CLINICAL TRIAL: NCT04746339
Title: Apixaban for PrOphyLaxis of thromboemboLic Outcomes in COVID-19 - the Apollo Trial
Brief Title: Apixaban for PrOphyLaxis of thromboemboLic Outcomes in COVID-19
Acronym: APOLLO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the decrease in COVID cases and in the recruitment rate, and DSMB orientation.
Sponsor: Brazilian Clinical Research Institute (Other)
Collaborators: Hospital Israelita Albert Einstein (Other); Hospital do Coracao (Other); Hospital Sirio-Libanes (Other); Hospital Moinhos de Vento (Other); Hospital Alemão Oswaldo Cruz (Other); Beneficência Portuguesa de São Paulo (Other); Brazilian Research In Intensive Care Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 004/2020
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Covid19; Thrombosis
Keywords: SARS-CoV2; Anticoagulation; Apixaban
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban Group (Active Comparator)
  Interventions: Drug: Apixaban 2.5 MG
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban 2.5 MG — Apixaban 2.5mg twice daily for 30 days
  Arms: Apixaban Group
Drug: Placebo — placebo twice daily for 30 days
  Arms: Placebo Group

SUMMARY:
Randomized, double-blinded, placebo-controlled trial comparing oral anticoagulation with placebo for community-dwelling patients with symptomatic COVID-19 infection and risk factors for thrombosis.

DETAILED DESCRIPTION:
Randomized, double-blinded, placebo-controlled trial comparing oral anticoagulation with placebo for community-dwelling patients with symptomatic COVID-19 infection and risk factors for thrombosis.

Randomization 1:1 - Group 1 will receive Apixaban 2.5mg twice daily vs. matching placebo (Group 2) for 30 days.

Primary Objective: To evaluate the clinical impact of a strategy of oral anticoagulation with apixaban comparing with placebo on the number of days alive and out of the hospital/emergency department (DAOH) through 30 days in outpatients with symptomatic SARS-CoV2 infection and risk factors for thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with symptomatic laboratory-proven diagnosis of COVID-19 (any exam that shows acute infection as positive PCR or IgM in a context of acute symptoms ≤ 10 days) AND
* Negative pregnancy test for women in child bearing period AND
* D-dimer level ≥ 2x ULN or
* C-reactive protein (CRP) ≥ 10 mg/L or
* At least two of the following risk factors:

  * d-dimer level ≥ULN
  * CRP ≥ULN
  * age ≥65,
  * diabetes,
  * chronic kidney disease stage 3
  * cardiopulmonary disease (for example, peripheral arterial disease, coronary artery disease, heart failure, chronic obstructive pulmonary disease),
  * history of PE/DVT,
  * nursing home/SNF resident or severely restricted mobility
  * Body mass index ≥30 kg/m2.

Exclusion Criteria:

* Age < 18 years-old
* Patients with indication for full anticoagulation during inclusion (for example, diagnosis of venous thromboembolism, atrial fibrillation, mechanical valve prosthesis)
* Platelets < 50,000 /mm3
* Use of acetylsalicylic acid > 100 mg per day
* Use of P2Y12 inhibitor (clopidogrel, prasugrel, ticagrelor)
* Chronic use of NSAIDs
* Hypersensitivity to apixaban
* Creatinine clearance < 30 ml/min
* Pregnancy or breastfeeding
* Patients contraindicated to anticoagulation (active bleeding, recent major surgery, blood dyscrasia or prohibitive hemorrhage risk as evaluated by the investigator)
* A history of hemorrhagic stroke or any intracranial bleeding at any time in the past or current intracranial neoplasm (benign or malignant), cerebral metastases, arteriovenous (AV) malformation, or aneurysm
* Use of strong inhibitors of cytochrome P450 (CYP) 3A4 and/or P-glycoprotein (P-gp) (e.g. protease inhibitors, ketoconazole, Itraconazole) and/or use of P-gp and strong CYP3A4 inducers (such as but not limited to rifampin/rifampicin, rifabutin, rifapentine, phenytoin, phenobarbital, carbamazepine, or St. John's Wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of days alive and out of hospital or emergency department | In 30 days
  Number of days alive and out of hospital or emergency department through 30 days.

SECONDARY OUTCOMES:
Hospitalization due to bleeding | In 30 days
Hospitalizations for cardiopulmonary causes | In 30 days
All-cause hospitalization | In 30 days
All-cause death | In 30 days
Days free of venous thromboembolism | In 30 days
  Venous thromboembolism (VTE) include deep venous thrombosis and pulmonary embolism.
Major cardiovascular events (MACE) | In 30 days
  Major cardiovascular events (MACE) includes cardiovascular death, myocardial infarction (MI) and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Renato D. Lopes, MD, PhD, Study Chair — BCRI
Locations (4):
- Brazil (4):
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Hospital Universitário São Francisco de Assis, Bragança Paulista, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital Santa Paula, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All data provided during study is anonymized to respect the privacy of patients who have participated in the trial in line with applicable regulations.

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523